CLINICAL TRIAL: NCT02529137
Title: Pivotal Study for Validation of Philips Dx for Diagnosis in Surgical Pathology
Brief Title: Pivotal Study for Validation of Philips Dx (PDx)
Status: Completed | Type: Observational
Sponsor: Philips Digital & Computational Pathology (Industry)
Responsible Party: Sponsor
Other Study IDs: DPS-CT-0007
Record Dates: First submitted 2015-08-18; First posted 2015-08-20 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Pathologic Processes
MeSH Terms: conditions — Pathologic Processes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical pathology cases: Cases will be selected from the sites Laboratory Information Systems using the in- and exclusion criteria.

SUMMARY:
The primary objective of this study is to show safety and effectiveness of the PDx for In Vitro Diagnostic (IVD) use as an aid to the pathologist to view, review and diagnose digital images of surgical pathology slides.

ELIGIBILITY:
Inclusion Criteria

* All relevant coverslipped slide or slides, with human tissue obtained via surgical pathology of original case are available.
* Original sign-out diagnosis is available.
* The selected slide or slides fulfill the quality checks according to general clinical practice.
* Target enrollment of organs and subtypes according pre-specified list.

Exclusion Criteria

* Cases, including sent out cases, for which any of the relevant slides used for the original sign-out diagnosis is no longer available at the site.
* The selected slide or slides do not match any subtype of the organ for which the case was selected.
* Relevant Clinical Information that was available to the sign-out pathologist in the pathology request form cannot be obtained.
* Selected slides contain indelible markings.
* Selected slides with damaged tissue.
* More than one case was selected for a patient (only one case may be enrolled per patient).
* Case consists of frozen section(s) only.
* Case consists of gross specimens only.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Both: surgical pathology slides of both female and male participants are being studied.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mischa Nelis, Study Director — Philips DPS
Locations (4):
- United States (4):
  - Shady Grove Adventist, Silver Spring, Maryland
  - Cleveland Clinic, Cleveland, Ohio
  - Miraca Life Sciences, Irving, Texas
  - University of Virginia, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Case enrollment started in October 2015 and enrollment was completed in December 2015. A total of 2000 cases was enrolled. Eight cases were discontinued before reading, resulting in a total of 1992 cases for reading.
Pre-assignment Details: In total 2000 cases were planned to be enrolled, divided over the clinical study sites.
  A total of 2000 cases were enrolled, between 390 and 600 cases per site over four sites.
Groups:
- Surgical Pathology Cases: Cases were selected from the sites Laboratory Information Systems using the in- and exclusion criteria. Each pathologist read the cases per block of 20 cases, alternating between Manual Optical and Manual Digital per block, i.e. all cases were evaluated by both modalities. At each site two pathologists were randomly assigned to the reading sequence starting with MO and two pathologists to the reading sequence starting with MD. There was no intervention in this study.
Period: Overall Study
Arm/Group | Surgical Pathology Cases
Started (Instead of participants, retrospective cases were enrolled in the study) | 2000
Completed (Instead of participants, retrospective cases were enrolled in the study) | 1992
Not Completed | 8
Not completed — Discontinuation for different reasons | 8

BASELINE CHARACTERISTICS:
Population: Surgical pathology cases where diagnosis was already rendered for more than one year before start of study
Units Other Than Participants: cases
Arm/Group | Surgical Pathology Cases
Number analyzed (Participants) | 2000
Number analyzed (cases) | 1992
Age, Categorical [Count of Units; unit: cases]
  <=18 years | NA — data were not collected
  Between 18 and 65 years | NA — data were not collected
  >=65 years | NA — data were not collected
Sex: Female, Male [Count of Units; unit: cases]
  Female | NA — data were not collected
  Male | NA — data were not collected
Region of Enrollment [Number; unit: cases]
  United States | 1992

OUTCOME MEASURES:

1. Primary Outcome: Major Discordance Rate
Description: The primary endpoint was the difference in major discordance rates between Manual Optical (MO) and Manual Digital (MD). MO is defined as reading by using optical microscope whereas MD is defined as reading by using PIPS. MO major discordance rate is defined as the proportion of major discordances between the MO diagnosis and the main diagnosis from the total number of readings.
  MD major discordance rate is defined as the proportion of major discordances between the MD diagnosis and the main diagnosis from the total number of readings.
Time Frame: 6 months
Population: 8 cases were discontinued for reasons such as broken/damaged slide (1), slide size did not meet the scanner specifications (4), no tissue detected by the scanner (2) and more than one case was selected for the patient (1).
Measure: Number (95% Confidence Interval); unit: percentage of major discordance
Units Other Than Participants: Readings
Groups:
- Manual Optical (MO): MO is defined as reading by using optical microscope. Reading results in a diagnosis. This diagnosis is later compared to the main diagnosis resulting in either concordance, minor discordance or major discordance.
- Manual Digital (MD): MD is defined as reading by using PIPS. Reading results in a diagnosis. This diagnosis is later compared to the main diagnosis resulting in either concordance, minor discordance or major discordance.
Arm/Group | Manual Optical (MO) | Manual Digital (MD)
Number analyzed (Participants) | 1992 | 1992
Number analyzed (Readings) | 7961 | 7964
percentage of major discordance | 4.4 [3.02 to 6.33] | 4.7 [3.27 to 6.82]
Statistical Analysis 1: Comparison: Manual Optical (MO) vs Manual Digital (MD); Test type: Non-Inferiority — the non-inferiority margin was set at 4%; difference = 0.4, 95% CI 2-sided [-0.30 to 1.01]

ADVERSE EVENTS:
Time Frame: From study start to study closure (11 months)
Arm/Group | Surgical Pathology Cases
All-Cause Mortality (participants affected / at risk) | 0/2000
Serious Adverse Events (participants affected / at risk) | 0/2000
Other Adverse Events (participants affected / at risk) | 0/2000

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less